CLINICAL TRIAL: NCT06649630
Title: Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Intravenous, Oral and Subcutaneous Doses of Inno8 in Healthy Male Participants
Brief Title: A Study Looking at How Different Doses of Study Medicine (Inno8) Works in the Body of Healthy Men
Acronym: VOYAGER1
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NN7442-7582; U1111-1292-7153 (Other: Universal Trial Number); 2023-506520-90 (Other: EU CT Number)
Record Dates: First submitted 2024-10-14; First posted 2024-10-21 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Haemophilia A
MeSH Terms: conditions — Hemophilia A

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Sponsor staff involved in the clinical trial is masked according to company standard procedures.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (14):
- Cohort 1 (SAD): NNC0442-0344 A (Experimental): Participants will receive single dose of NNC0442-0344 A intravenously.
  Interventions: Drug: NNC0442-0344 A
- Cohort 2 (SAD): NNC0442-0344 A (Experimental): Participants will receive single dose of NNC0442-0344 A intravenously.
  Interventions: Drug: NNC0442-0344 A
- Cohort 3 (SAD): NNC0442-0344 A (Experimental): Participants will receive single dose of NNC0442-0344 A intravenously.
  Interventions: Drug: NNC0442-0344 A
- Cohort 4 (SAD): NNC0442-0344 A (Experimental): Participants will receive single dose of NNC0442-0344 A intravenously.
  Interventions: Drug: NNC0442-0344 A
- Cohort 5 (SAD): NNC0442-0344 A (Experimental): Participants will receive single dose of NNC0442-0344 A intravenously.
  Interventions: Drug: NNC0442-0344 A
- Cohort 1 (MAD): NNC0442-0344 A (Experimental): Participants will receive a oral daily dose of NNC0442-0344 A for 10 days.
  Interventions: Drug: NNC0442-0344 A
- Cohort 2 (MAD): NNC0442-0344 A (Experimental): Participants will receive a oral daily dose of NNC0442-0344 A for 10 days.
  Interventions: Drug: NNC0442-0344 A
- Cohort 3 (MAD): NNC0442-0344 A (Experimental): Participants will receive a oral daily dose of NNC0442-0344 A for 10 days.
  Interventions: Drug: NNC0442-0344 A
- Cohort 4 (MAD): NNC0442-0344 A (Experimental): Participants will receive a oral daily dose of NNC0442-0344 A for 10 days.
  Interventions: Drug: NNC0442-0344 A
- Cohort 1 (SSD): NNC0442-0344 A (Experimental): Participants will receive single dose of NNC0442-0344 A subcutaneously.
  Interventions: Drug: NNC0442-0344 A
- Cohort 2 (SSD): NNC0442-0344 A (Experimental): Participants will receive single dose of NNC0442-0344 A subcutaneously.
  Interventions: Drug: NNC0442-0344 A
- SAD: Placebo (Placebo Comparator): Participants will receive single dose of placebo intravenously.
  Interventions: Drug: Placebo
- MAD: Placebo (Placebo Comparator): Participants will receive a oral daily dose of Placebo for 10 days.
  Interventions: Drug: Placebo
- SSD: Placebo (Placebo Comparator): Participants will receive single dose of placebo subcutaneously.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: NNC0442-0344 A — SAD: NNC0442-0344 A will be administered intravenously.
  MAD: NNC0442-0344 A will be administered orally.
  SSD: NNC0442-0344 A will be administered subcutaneously.
  Other Names: Inno8
  Arms: Cohort 1 (MAD): NNC0442-0344 A; Cohort 1 (SAD): NNC0442-0344 A; Cohort 1 (SSD): NNC0442-0344 A; Cohort 2 (MAD): NNC0442-0344 A; Cohort 2 (SAD): NNC0442-0344 A; Cohort 2 (SSD): NNC0442-0344 A; Cohort 3 (MAD): NNC0442-0344 A; Cohort 3 (SAD): NNC0442-0344 A; Cohort 4 (MAD): NNC0442-0344 A; Cohort 4 (SAD): NNC0442-0344 A; Cohort 5 (SAD): NNC0442-0344 A
Drug: Placebo — SAD: Placebo will be administered intravenously.
  MAD: Placebo will be administered orally.
  SSD: Placebo will be administered subcutaneously.
  Arms: MAD: Placebo; SAD: Placebo; SSD: Placebo

SUMMARY:
This study will test how different doses of study medicine (Inno8) work in the healthy men. The purpose of this study is to prove safety of Inno8 in healthy men, which will support further development of Inno8 in people with Haemophilia A. The study consists of three parts: single ascending dose (SAD), multiple ascending dose (MAD) and single subcutaneous dose (SSD). Each part will have more than one cohort (like sub-parts). No matter which part the participants will be enrolled in, they will either get the study medicine (Inno8) or a dummy medicine that looks like the study medicine but has no effect on the body (placebo). Which treatment participants get is decided by chance. The study medicine is a new medicine that cannot be prescribed by doctors. In the SAD and SSD part participants will receive a single injection of study medicine or placebo, and the study will last for up to 9 weeks. In the MAD part, participants will receive 1-2 tablets of study medicine or placebo daily for 10 days, and the study will last for up to 11 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Age 18-45 years (both inclusive) at the time of signing informed consent
* Body mass index between 18.5 and 29.9 Kilogram Per Square Meter (kg/m^2) (both inclusive)
* Body weight between 60.0 and 100.0 Kilogram (kg) (both inclusive)
* Considered to be generally healthy based on the medical history, physical examination, and the results of vital signs, electrocardiogram and clinical laboratory tests performed during the screening visit, as judged by the investigator

Exclusion Criteria:

* Factor VIII activity greater than or equal to (≥) 150% at screening
* Increased risk of thrombosis, e.g. known history of personal or first-degree relative(s) with unprovoked deep vein thrombosis
* Any clinical signs or established diagnosis of venous or arterial thromboembolic disease
* Any of the thrombophilia markers listed below:
* Protein C, protein S or antithrombin below the lower normal laboratory range
* Factor II activity, activated protein C resistance, lupus anticoagulant, anti-cardiolipin antibody (IgG and IgM) or anti-β2 glycoprotein I antibody (IgG and IgM) outside the normal laboratory range at screening

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 108 (Estimated)
Dates: Start 2024-09-23 (Actual); Primary Completion 2026-05-04 (Estimated); Study Completion 2026-05-04 (Estimated)

PRIMARY OUTCOMES:
SAD: Number of treatment emergent adverse events | From time of dosing (Day 1) to Day 36
  Measured as count of events.
MAD: Number of treatment emergent adverse events | From time of dosing (Day 1) to end of follow-up (Day 46)
  Measured as count of events.
SSD: Number of treatment emergent adverse events | From time of dosing (Day 1) to Day 36
  Measured as count of events.

SECONDARY OUTCOMES:
SAD: Change in D-dimer | From baseline (Day 1) to Day 36
  Measured as absolute and percentage (%).
SAD: Change in prothrombin fragment 1 and 2 | From baseline (Day 1) to Day 36
  Measured as absolute and %.
SAD: Change in fibrinogen | From baseline (Day 1) to Day 36
  Measured as absolute and %.
SAD: Change in platelets | From baseline (Day 1) to Day 36
  Measured as absolute and %.
SAD: Cmax, SD: the maximal concentration of Inno8 after a single dose | From baseline (Day 1) to Day 36
  Measured as nanograms per millilitre (ng/mL).
SAD: AUC, SD: the area under the concentration curve of Inno8 after a single dose | From baseline (Day 1) to Day 36
  Measured as nanograms*day per millilitre (ng*day/mL).
SAD: T1/2, SD: the terminal half-life of Inno8 after a single dose | From baseline (Day 1) to Day 36
  Measured as days.
SAD: Maximum change in activated partial thromboplastin time | From baseline (Day 1) to Day 36
  Measured as seconds.
SAD: Maximum thrombin generation (peak height) | From baseline (Day 1) to Day 36
  Measured as nanomolar (nM).
MAD: Change in D-dimer | From baseline (Day 1) to Day 46
  Measured as absolute and %.
MAD: Change in prothrombin fragment 1 and 2 | From baseline (Day 1) to Day 46
  Measured as absolute and %.
MAD: Change in fibrinogen | From baseline (Day 1) to Day 46
  Measured as absolute and %.
MAD: Change in platelets | From baseline (Day 1) to Day 46
  Measured as absolute and %.
MAD: Occurrence of anti-Inno8 antibodies | From baseline (Day 1) to Day 46
  Measured as count.
MAD: Cmax: The maximum concentration of Inno8 after multiple doses | From Day 10 to Day 11
  Measured as ng/mL.
MAD: Tmax: The time to Cmax after last multiple dose | From Day 10 to Day 11
  Measured as hours.
MAD: Tmax: The time to Cmax after first dose | From Day 1 to Day 2
  Measured as hours.
MAD: AUC: the area under the Inno8 concentration-time curve in the dosing interval after multiple doses | From Day 10 to Day 11
  Measured as ng*day/mL.
MAD: Maximum thrombin generation (peak height) | From Day 10 to Day 11
  Measured as nM.
SSD: Change in D-dimer | From baseline (Day 1) to Day 36
  Measured as absolute and %.
SSD: Change in prothrombin fragment 1 and 2 | From baseline (Day 1) to Day 36
  Measured as absolute and %.
SSD: Change in fibrinogen | From baseline (Day 1) to Day 36
  Measured as absolute and %.
SSD: Change in platelets | From baseline (Day 1) to Day 36
  Measured as absolute and %.
SSD: Cmax, SD: the maximal concentration of Inno8 after a single dose | From baseline (Day 1) to Day 36
  Measured as ng/mL.
SSD: AUC, SD: the area under the concentration curve of Inno8 after a single dose | From baseline (Day 1) to Day 36
  Measured as ng*day/mL.
SSD: T1/2, SD: the terminal half-life of Inno8 after a single dose | From baseline (Day 1) to Day 36
  Measured as days.
SSD: Maximum change in activated partial thromboplastin time | From baseline (Day 1) to Day 36
  Measured as seconds.
SSD: Maximum thrombin generation (peak height) | From baseline (Day 1) to Day 36
  Measured as nanomolar (nM).

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 2834), Study Director — Novo Nordisk A/S
Locations (2):
- Germany (2):
  - Charité - Campus Charité Mitte - Charité Research Organisation GmbH, Berlin
  - Charité Research Organisation GmbH, Berlin

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: https://novonordisk-trials.com